CLINICAL TRIAL: NCT00891462
Title: Efficacy and Safety of Aclidinium Bromide at Two Dose Levels (200 μg Twice Daily, 400 μg Twice Daily) vs. Placebo When Administered to Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety of Aclidinium Bromide for Treatment of Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD) (LAS-MD-33)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAS-MD-33; ACCORD COPD I
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis; Emphysema; Airflow Obstruction, Chronic; Chronic Airflow Obstruction; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Aclidinium bromide dose, inhaled, for 12 weeks of treatment
  Interventions: Drug: Aclidinium bromide
- 2 (Experimental): Aclidinium bromide dose, inhaled, for 12 weeks of treatment
  Interventions: Drug: Aclidinium bromide
- 3 (Placebo Comparator): Inhaled placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide — Aclidinium bromide 200 μg, oral inhalation twice per day for 12 weeks of treatment
  Arms: 1
Drug: Aclidinium bromide — Aclidinium bromide 400 μg, oral inhalation twice per day for 12 weeks of treatment
  Arms: 2
Drug: Placebo — Dose-matched placebo, oral inhalation twice per day for 12 weeks of treatment
  Arms: 3

SUMMARY:
The purpose of this study is to assess the efficacy (effectiveness) and safety of aclidinium bromide doses as compared to placebo in the treatment of moderate to severe chronic obstructive pulmonary disease. The study will be 16 weeks in duration; 2-week run-in period, 12-week double-blind treatment, and 2-week follow-up phone visit.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of stable moderate to severe COPD as defined by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, 2009; postbronchodilator FEV1/FVC < 70%, and postbronchodilator FEV1 ≥ 30% and < 80% predicted
* Current or former cigarette smokers

Exclusion Criteria:

* Patients who have been hospitalized for an acute COPD exacerbation within 3 months before the first visit
* Respiratory tract infection or COPD exacerbation in the 6 weeks before Visit 1
* Patient with any clinically significant respiratory conditions other than COPD, cardiovascular conditions or mental illness
* History or presence of asthma verified from medical records
* Chronic use of oxygen therapy greater than or equal to 15 hours per day
* Patient with uncontrolled infection due to HIV and/or active hepatitis
* Patients with a history of hypersensitivity reaction to inhaled anticholinergics
* Patients with clinically significant cardiovascular conditions, including myocardial infarction during the previous 6 months, newly diagnosed arrhythmia within the previous 3 months, unstable angina, unstable arrhythmia that had required changes in pharmacological therapy or other intervention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (100):
- United States (93):
  - Forest Investigative Site, Birmingham, Alabama
  - Forest Investigative Site, Jasper, Alabama
  - Forest Investigative Site, Mobile, Alabama
  - Forest Investigative Site, Mesa, Arizona
  - Forest Investigative Site, Phoenix, Arizona
  - Forest Investigative Site, Anaheim, California
  - Forest Investigative Site, Encinitas, California
  - Forest Investigative Site, Fresno, California
  - Forest Investigative Site, Fullerton, California
  - Forest Investigative Site, Lakewood, California
  - Forest Investigative Site, Orange, California
  - Forest Investigative Site, Palo Alto, California
  - Forest Investigative Site, Rancho Mirage, California
  - Forest Investigative Site, Sacramento, California
  - Forest Investigative Site, San Diego, California
  - Forest Investigative Site, Colorado Springs, Colorado
  - Forest Investigative Site, Denver, Colorado
  - Forest Investigative Site, Wheat Ridge, Colorado
  - Forest Investigative Site, Waterbury, Connecticut
  - Forest Investigative Site, Brandon, Florida
  - Forest Investigative Site, Clearwater, Florida
  - Forest Investigative Site, DeLand, Florida
  - Forest Investigative Site, Fort Lauderdale, Florida
  - Forest Investigative Site, Melbourne, Florida
  - Forest Investigative Site, Ormond Beach, Florida
  - Forest Investigative Site, Panama City, Florida
  - Forest Investigative Site, Pensacola, Florida
  - Forest Investigative Site, Tamarac, Florida
  - Forest Investigative Site, Tampa, Florida
  - Forest Investigative Site, Austell, Georgia
  - Forest Investigative Site, Blue Ridge, Georgia
  - Forest Investigative Site, Duluth, Georgia
  - Forest Investigative Site, Marietta, Georgia
  - Forest Investigative Site, River Forest, Illinois
  - Forest Investigative Site, Skokie, Illinois
  - Forest Investigative Site, South Bend, Indiana
  - Forest Investigative Site, Crescent Springs, Kentucky
  - Forest Investigative Site, Lexington, Kentucky
  - Forest Investigative Site, Lafayette, Louisiana
  - Forest Investigative Site, Bangor, Maine
  - Forest Investigative Site, Baltimore, Maryland
  - Forest Investigative Site, Hagerstown, Maryland
  - Forest Investigative Site, North Dartmouth, Massachusetts
  - Forest Investigative Site, Livonia, Michigan
  - Forest Investigative Site, Edina, Minnesota
  - Forest Investigative Site, Minneapolis, Minnesota
  - Forest Investigative Site, Florissant, Missouri
  - Forest Investigative Site, Saint Charles, Missouri
  - Forest Investigative Site, Billings, Montana
  - Forest Investigative Site, Butte, Montana
  - Forest Investigative Site, Papillion, Nebraska
  - Forest Investigative Site, Berlin, New Jersey
  - Forest Investigative Site, Summit, New Jersey
  - Forest Investigative Site, Brooklyn, New York
  - Forest Investigative Site, Buffalo, New York
  - Forest Investigative Site, Great Neck, New York
  - Forest Investigative Site, Ithaca, New York
  - Forest Investigative Site, New Hyde Park, New York
  - Forest Investigative Site, New York, New York
  - Forest Investigative Site, Asheville, North Carolina
  - Forest Investigative Site, Charlotte, North Carolina
  - Forest Investigative Site, Raleigh, North Carolina
  - Forest Investigative Site, Canton, Ohio
  - Forest Investigative Site, Cincinnati, Ohio
  - Forest Investigative Site, Columbus, Ohio
  - Forest Investigative Site, Toledo, Ohio
  - Forest Investigative Site, Oklahoma City, Oklahoma
  - Forest Investigative Site, Medford, Oregon
  - Forest Investigative Site, Portland, Oregon
  - Forest Investigative Site, Bethlehem, Pennsylvania
  - Forest Investigative Site, Erie, Pennsylvania
  - Forest Investigative Site, Hershey, Pennsylvania
  - Forest Investigative Site, Pittsburgh, Pennsylvania
  - Forest Investigative Site, Upland, Pennsylvania
  - Forest Investigative Site, East Providence, Rhode Island
  - Forest Investigative Site, Johnston, Rhode Island
  - Forest Investigative Site, Charleston, South Carolina
  - Forest Investigative Site, Greenville, South Carolina
  - Forest Investigative Site, Greer, South Carolina
  - Forest Investigative Site, Spartanburg, South Carolina
  - Forest Investigative Site, Nashville, Tennessee
  - Forest Investigative Site, Dallas, Texas
  - Forest Investigative Site, Fort Worth, Texas
  - Forest Investigative Site, Houston, Texas
  - Forest Investigative Site, San Antonio, Texas
  - Forest Investigative Site, Tyler, Texas
  - Forest Investigative Site, Waco, Texas
  - Forest Investigative Site, Midvale, Utah
  - Forest Investigative Site, Richmond, Virginia
  - Forest Investigative Site, Bellingham, Washington
  - Forest Investigative Site, Spokane, Washington
  - Forest Investigative Site, Tacoma, Washington
  - Forest Investigative Site, Milwaukee, Wisconsin
- Canada (7):
  - Forest Investigative Site, Saskatoon, Saskatchewan
  - Forest Investigative Site, Edmonton
  - Forest Investigative Site, Hamilton
  - Forest Investigative Site, Kelowna
  - Forest Investigative Site, Niagara Falls
  - Forest Investigative Site, Sainte-Foy
  - Forest Investigative Site, Toronto

REFERENCES:
- [Derived] McGarvey L, Morice AH, Smith JA, Birring SS, Chuecos F, Seoane B, Jarreta D. Effect of aclidinium bromide on cough and sputum symptoms in moderate-to-severe COPD in three phase III trials. BMJ Open Respir Res. 2016 Dec 8;3(1):e000148. doi: 10.1136/bmjresp-2016-000148. eCollection 2016. PMID 28074135
- [Derived] Kerwin EM, D'Urzo AD, Gelb AF, Lakkis H, Garcia Gil E, Caracta CF; ACCORD I study investigators. Efficacy and safety of a 12-week treatment with twice-daily aclidinium bromide in COPD patients (ACCORD COPD I). COPD. 2012 Apr;9(2):90-101. doi: 10.3109/15412555.2012.661492. Epub 2012 Feb 9. PMID 22320148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred from April to July of 2009 at 106 study sites, (100 in the United States and 6 additional sites in Canada.) A total of 99 study sites randomized patients.
Pre-assignment Details: From the total of 561 patients randomized, 560 patients received at least 1 dose of double-blind treatment and therefore were included in the Safety Population. Of these patients, 559 had at least 1 postbaseline FEV1 assessment and qualified for the Intent to Treat (ITT) Population.
Groups:
- Placebo: Inhaled placebo for 12 weeks
- Aclidinium Bromide, 200µg: Aclidinium bromide, 200 microgram dose. Oral inhalation, twice per day, for 12 weeks of treatment
- Aclidinium Bromide, 400µg: Aclidinium bromide 400 microgram dose. Oral inhalation, twice per day, for 12 weeks of treatment.
Period: Overall Study
Arm/Group | Placebo | Aclidinium Bromide, 200µg | Aclidinium Bromide, 400µg
Started | 186 | 185 | 190
Completed | 149 | 152 | 166
Not Completed | 37 | 33 | 24
Not completed — Withdrawal by Subject | 9 | 6 | 7
Not completed — Adverse Event | 7 | 8 | 7
Not completed — Lack of Efficacy | 10 | 5 | 1
Not completed — COPD exacerbation | 7 | 4 | 1
Not completed — Other Reason | 2 | 5 | 3
Not completed — Protocol Violation | 2 | 1 | 3
Not completed — Inclusion/exclusion criteria | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aclidinium Bromide, 200µg | Aclidinium Bromide, 400µg | Total
Number analyzed (Participants) | 186 | 184 | 190 | 560
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (9.2) | 63.1 (9.5) | 64.9 (9.5) | 64.3 (9.4)
Age, Customized [Number; unit: participants]
  ≥ 40 to < 60 years | 46 | 64 | 44 | 154
  ≥ 60 to < 70 years | 85 | 72 | 87 | 244
  ≥ 70 years | 55 | 48 | 59 | 162
Gender [Count of Participants; unit: Participants]
  Female | 90 | 83 | 90 | 263
  Male | 96 | 101 | 100 | 297
Region of Enrollment [Number; unit: participants]
  United States | 176 | 170 | 177 | 523
  Canada | 10 | 14 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose Forced Expiratory Volume in 1 Second (FEV1)
Description: Change from baseline in trough forced expiratory volume in 1 second before the morning dose of aclidinium bromide, Last Observation Carried Forward (LOCF)
Time Frame: Change from Baseline to 12 weeks
Population: Of 561 patients randomized, 560 patients received at least 1 dose of double-blind treatment and therefore were included in the Safety Population. Of these patients, 559 had a baseline and at least 1 postbaseline FEV1 assessment and qualified for the Intent to Treat (ITT) Population. The primary efficacy endpoint was based on ITT population.
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- Placebo: Dose-matched placebo twice per day, inhaled for 12 weeks of treatment
Arm/Group | Placebo | Aclidinium Bromide, 200µg | Aclidinium Bromide, 400µg
Number analyzed (Participants) | 185 | 184 | 190
L | -0.025 (0.015) | 0.062 (0.015) | 0.099 (0.015)
Statistical Analysis 1: Comparison: Placebo vs Aclidinium Bromide, 200µg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = 0.086, 95% CI 2-sided [0.05 to 0.13]
Statistical Analysis 2: Comparison: Placebo vs Aclidinium Bromide, 400µg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = 0.124, 95% CI 2-sided [0.08 to 0.16]

2. Secondary Outcome: Change From Baseline in Peak Forced Expiratory Volume in 1 Second (FEV1)
Description: Change From Baseline in Peak FEV1 (L) at Week 12, Last Observation Carried Forward (LOCF)
Time Frame: Change from Baseline to 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- Placebo: Dose matched placebo twice per day, inhaled for 12 weeks of treatment
- Aclidinium Bromide, 200 µg: Aclidinium bromide, 200 µg dose, Oral inhalation, twice per day, for 12 weeks of treatment
Arm/Group | Placebo | Aclidinium Bromide, 200 µg | Aclidinium Bromide, 400µg
Number analyzed (Participants) | 185 | 184 | 190
L | 0.071 (0.016) | 0.217 (0.016) | 0.263 (0.016)

ADVERSE EVENTS:
Time Frame: Adverse events reporting occurred from April 28th, 2009 to December 3rd, 2009 at 99 study sites.
Arm/Group | Placebo | Aclidinium Bromide, 200µg | Aclidinium Bromide, 400µg
Serious Adverse Events (participants affected / at risk) | 4/186 | 8/184 | 6/190
Other Adverse Events (participants affected / at risk) | 23/186 | 17/184 | 14/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Aclidinium Bromide, 200µg (N=184) | Aclidinium Bromide, 400µg (N=190)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 2 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Aclidinium Bromide, 200µg (N=184) | Aclidinium Bromide, 400µg (N=190)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 | 17 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute.